CLINICAL TRIAL: NCT05895526
Title: Comparison of the Clinical Effectiveness of Self Etch Adhesive and Fluoride Varnish in Reducing Dentin Hypersensitivity in Patients With Gingival Recession: Randomized Clinical Trial
Brief Title: Comparison of the Effectiveness of Self Etch Adhesive and Fluoride Varnish in Reducing Hypersensitivity in Patients With Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prime Foundation (Other)
Responsible Party: Principal Investigator, Iftikhar Akbar, Professor, Prime Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDC
Record Dates: First submitted 2023-04-12; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Dentin Sensitivity
Keywords: Dentin permeability; Dentin hypersensitivity; Gingival recession
MeSH Terms: conditions — Dentin Sensitivity; Gingival Recession

STUDY DESIGN:
Intervention Model Description: 1. Group A (Application of 5% sodium fluoride varnish)
  2. Group B (Self etch dentin adhesive)
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% Sodium Fluoride Varnish (Experimental): 71 patients will be in 5% Sodium Fluoride Varnish
  Interventions: Procedure: Self etch dentin adhesive, Fluoride varnish
- Self Etch Dentin Adhesive (Experimental): 71 patients will be in Self Etch Dentin Adhesive
  Interventions: Procedure: Self etch dentin adhesive, Fluoride varnish

INTERVENTIONS:
Procedure: Self etch dentin adhesive, Fluoride varnish — After an informed consent, in one group 5% sodium fluoride varnish will be applied in affected area, while the other group will receive self etch dentin adhesive.

SUMMARY:
Comparison of the clinical effectiveness of self etch adhesive and fluoride varnish in reducing dentin hypersensitivity in patients with gingival recession. A Randomized Clinical Trial

ABSTRACT Objective: To compare the clinical effectiveness of self etch adhesive and fluoride varnish in reducing dentin hypersensitivity in patients with gingival recession

Study Design: Randomized Clinical Trial Place of Study: Department of Operative Dentistry and Endodontics, Peshawar Dental College, Warsak Road.

Methodology: 142 diagnosed cases of Dentin hypersensitivity from outpatient department of nephrology, Prime Hospital Peshawar will be referred to operative department, Peshawar dental college for Comparison of the clinical effectiveness of self etch adhesive and fluoride varnish in reducing dentin hypersensitivity in patients with gingival recession.

Results:

Conclusion:

DETAILED DESCRIPTION:
Dentin hypersensitivity is a common disorder and is one of the most irritating clinical condition1. It is one of the everyday complaints from patient visiting dental operatory2. Dentin hypersensitivity has been defined as "Short, sharp pain arising from exposed dentin in response to stimuli typically thermal, evaporative , tactile , osmotic or chemical that cannot be related to any other dental defect or pathology"3'4.Prevalance of dentin hypersensitivity in general population is 4% to 57% 5. Adults are normally affected by dentin hypersensitivity mainly in their late 30s however mainly people aged between 29 to 49 years can also suffer from this6.

One of the most well known theory for dentin hypersensitivity is Brannstorm and Astrom's Hydrodynamic theory2'6. According to this theory environmental ,thermal, chemical changes cause the movement of fluid within tubules, which stimulate terminals of pulpal nerve fibers located in tubules, this will lead to acute transient pain6'7.

Dentin is composed of dentinal tubules and dentin is protected by highly mineralized structures i.e enamel covers the dentin in crown portion while root dentin is protected by cementum8.Certain type of physical, chemical, pathological and biological challenges or developing defects can lead to exposure of dentin. Periodontal tissue loss or gingival recession is one of the most predisposing factor because it will lead to exposure of cervical and root dentin2.

A lot of research has been done on treatment of dentin hypersensitivity but still no consensus has been reached on which product is "gold standard" for treatment of dentin hypersensitivity9.Lukomsky suggested that fluoride can be used as topical desensitizing agent for reduction of DH. It has been in use since 1941.Fluoride causes formation of calcium fluoride crystals and varying degree of fluorapatite which will block the transmission of noxious stimuli to pulp. For treatment of dentin hypersensitivity varnishes containing sodium fluoride as an active component are in use for many years9.Some researchers recommended the use of self etch adhesive for reduction of dentin permeability10.Self etch adhesive form acid resistant hybrid layer due to which they show high level of clinical effectiveness. Yu et al showed that one bottle self etch adhesive plays an effective role in alleviating symptoms of dentin hypersensitivity11.

The aim of current clinical study is to compare clinical effectiveness of self etch and fluoride varnish in reducing dentin hypersensitivity in patients with gingival recession.

Approval to carry out the study was sought from institutional Ethical Review Committee at Peshawar dental college before start of study. Study design was randomized control trial. By using Open epi, the total sample size will be 142 by using a duration of hypersensitivity(pain score) in group A (1.79±1.47) while in group B (2.41±1.22) from a previous study of Ammarah Afreen by keeping 80% Power of the test and 95% confidence interval9.

A prospective randomized clinical study will be planned at Operative Dentistry and Endodontics Department from 12 June, 2023 to 12 ,August 2023.This single center, double blind prospective RCT study will be conducted in Peshawar Dental College and Hospital. The inclusion criteria will be dentin hypersensitivity due to Miller's Class 1 gingival recession, aged between 20-45yrs, without root filled teeth and the patients who are willing to participate in the study. Whereas pregnant and lactating mother, crowned teeth with extensive gingival recession and with cervical restoration will be excluded.

All the selected patients have Miller's Class1 gingival recession in which marginal tissue recession does not extend to the mucogingival junction. Patients were informed regarding purpose, procedure, risk and benefits of the study. Verbal and written informed consent was obtained from all patient regarding his/her participation in study, and they were assured of maintaining confidentiality of the data collected from them. A structured customized performa was specifically designed to record the findings of study. The subjects were randomized by using random number table to minimize bias.

Patients were divided into two groups. The Group 1(Control Group) received the treatment that was based on the fluoride varnish company's instruction whereas Group 2 patients were under treatment regimens based on self etch dentin adhesive company's instruction.Teeth that are hypersensitive were identified using straight probe running cervically evaluating each tooth response. Tooth response to cold air was assessed using standard air syringe of dental unit for one to two seconds. In Group 1, After baseline assessment hypersensitivity were cleaned with cotton pellet soaked in distilled water, fluoride varnish was applied according to company's instruction whereas in group 2 self-etch adhesive, Optibond TM was applied for 20 seconds, dried with high pressure air flow for 5 seconds and light cured for 10 seconds according to manufacturer instruction. All subjects were instructed not to brush their teeth, eat, drink or rinse their mouth for at least two hours after each treatment.

A clinical evaluation of each tooth was assessed by another investigator who was not involved with the treatment procedure. Air stimulation response measurement was done via VAS as the baseline evaluation (T0) before intervention and data was collected, on the day of intervention after application of agents(T1), after one week (T2) and one month after treatment (T3) using tactile and air blast stimuli. The same examiner calculated the total VAS score of each study group at each follow up time from the mean of VAS scores of all treated teeth of every subject in the same group.

Baseline characteristics will also be compared. SPSS 22(SPSS Inc, Chicago, IL) will be used for all statistical analyses. The independent sample t-test will be used to analyze samples. The chi-square test will be used to assess the differences between categoric variables. The comparisons will be considered statistically significant at P < .05.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with dentin hypersensitivity due to gingival recession.
2. Patients having Miller's Class 1 gingival recession.
3. Patient aged between 20-45yrs with gingival recession without other periodontal issues.
4. Patient without root filled teeth.
5. Patients who are willing to participate in the study.

Exclusion Criteria:

1. Teeth with extensive gingival recession.
2. Teeth with cervical restoration.
3. Pregnant and lactating mother.
4. Crowned teeth.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-06-12 (Estimated); Primary Completion 2023-08-12 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the clinical effectiveness of self etch adhesive and fluoride varnish in reducing dentin hypersensitivity in patients with gingival recession. A Randomized Clinical Trial | Two months
  Patients will be divided into two groups. The Group 1 will receive the treatment that is based on the fluoride varnish company's instruction whereas Group 2 patients will under treatment regimens based on self etch dentin adhesive company's instructions.A clinical evaluation of each tooth will be done by another investigator who will not be involved with the treatment procedure. Air stimulation response measurement will be done via Visual analogue scale with score 0( No pain) ,1 2 3 ( Mild pain) , 4 5 6 (Moderate Pain) , 7 8 9 10 (Severe pain).The baseline evaluation (T0) before intervention , on the day of intervention after application of agents(T1), after one week (T2) and one month after treatment (T3) using tactile and air blast stimuli.The same examiner will calculate the total Visual analogue scale score of each study group at each follow up time from the mean of Visual analogue scale scores of all treated teeth of every subject in the same group..

CONTACTS AND LOCATIONS:
Overall Officials: Rizwan Qureshi, BDS, FCPS, Study Chair — Peshawar Dental College
Locations (1):
- Peshawar Dental College, Peshawar, Khyber Pakhtunkhwa, Pakistan